CLINICAL TRIAL: NCT00093782
Title: A Phase II Study of CCI-779 in Metastatic Neuroendocrine Carcinomas
Brief Title: Temsirolimus in Treating Patients With Metastatic Neuroendocrine Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03053; PHL-021; 6171; N01CM17105 (NIH); N01CM17107 (NIH); N01CM17102 (NIH)
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2016-12

CONDITIONS: Metastatic Gastrointestinal Carcinoid Tumor; Pulmonary Carcinoid Tumor; Recurrent Gastrointestinal Carcinoid Tumor; Recurrent Islet Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Islet Cell | interventions — temsirolimus; Sirolimus

ARMS (1):
- Treatment (temsirolimus) (Experimental): Patients receive CCI-779 IV over 30 minutes on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve a CR or PR receive 2 additional courses beyond CR or PR.
  Interventions: Drug: temsirolimus; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: temsirolimus — Given IV
  Other Names: CCI-779; cell cycle inhibitor 779; Torisel
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well CCI-779 works in treating patients with progressive metastatic neuroendocrine tumors. Drugs used in chemotherapy, such as CCI-779, work in different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To assess the objective tumor response rate (i.e. partial or complete responses as defined by the RECIST criteria) in patients with progressive metastatic neuroendocrine tumours given CCI-779.

II. To assess the stable disease rate and duration, time to progression, median survival time, 1-year survival rate and toxicity in patients with metastatic neuroendocrine carcinomas given CCI-779. As of 19 July 2010, overall survival follow-up is to be discontinued for the four remaining patients on long term follow-up. At that point in time, these patients had been off-treatment for 3 to 5 years. Time to progression and median survival times will be based on the currently available data.

III. To measure baseline levels of various elements up- and downstream of the mammalian target of rapamycin (mTOR). Where post-treatment biopsies are available, they will be analyzed for suppression of elements in the mTOR pathway as well as for any effect on cell cycle progression, apoptosis or anti-angiogenic effects.

OUTLINE: This is an open-label, multicenter study.

Patients receive CCI-779 IV over 30 minutes on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve a complete response (CR) or partial response (PR) receive 2 additional courses beyond CR or PR.

Patients are followed up for survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed neuroendocrine tumours either of carcinoid histology or a carcinoma of pancreatic islet cell origin; small cell variant, endocrine organ carcinomas, and adrenal gland malignancies (including paragangliomas) are excluded from this study
* Patients must have progressive metastatic disease defined by one of the following occurring within 6 months of study entry:

  * At least a 25% increase in radiologically or clinically measurable disease
  * Appearance of any new lesion or
  * Deterioration in clinical status
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan
* Previous local therapy (e.g. chemoembolization or bland embolization) allowed if completed > 6 weeks prior to study entry; for patients who received local therapy prior to study entry, there must be either progression of measurable disease documented within the treatment field, or must have measurable disease outside the treatment field prior to study entry
* Previous chemotherapy, investigational agents or radioactive therapies (e.g. radioactive octreotide) allowed if completed > 4 weeks prior to study entry (> 6 weeks if last regimen contained BCNU or mitomycin C); for patients who received systemic therapy prior to study entry, there must be documented progression of measurable disease prior to study entry
* Patients must not have disease that is currently amenable to surgery; prior surgery is allowed no less than 6 weeks prior to study entry
* Previous radiation therapy is allowed if > 4 weeks have elapsed since delivery of a dose likely to have myelotoxic effects (e.g. ≥ 3000cGy to fields including substantial marrow)
* Life expectancy of greater than 3 months
* ECOG performance status ≤ 2 (Karnofsky ≥ 60%)
* Leukocytes ≥ 3.0 x 10^9/L
* Absolute neutrophil count ≥ 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Total bilirubin ≤ 1.25 x ULN
* AST(SGOT)/ALT(SGPT) ≤ 3 x ULN; < 5 x ULN with liver metastases
* Creatinine ≤ 1.5 x ULN OR creatinine clearance (CrCl) calculated ≥ 60mL/min/1.73m^2
* Fasting serum cholesterol =< 350 mg/dL (9.0 mmol/L)
* Triglycerides =< 400 mg/dL (4.56 mmol/L)
* Must be willing and able to undergo tumor biopsy once before and once during experimental therapy; patients must have tumor lesions accessible for biopsy for correlative studies; in cases where there is a medical contraindication to tumor biopsy, exception may be granted upon discussion with the Principal Investigator/Chair
* The effects of CCI-779 on the developing human fetus at the recommended therapeutic dose are unknown; for this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents concurrently or within 4 weeks of study entry
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to CCI-779
* Concurrent cancer from another primary site requiring treatment of any kind within the past 3 years; curatively treated non-melanoma skin cancer or in situ carcinoma of the cervix are allowed
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because CCI-779 is an inhibitor of mRNA translation with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with CCI-779, breastfeeding should be discontinued if the mother is treated with CCI-779
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with CCI-779; appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2003-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, Principal Investigator — Princess Margaret Hospital Phase 2 Consortium
Locations (1):
- Princess Margaret Hospital Phase 2 Consortium, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Temsirolimus)
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Number of participants accrued
Arm/Group | Treatment (Temsirolimus)
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 8
Age, Continuous [Median (Full Range); unit: years] | 58 [36 to 78]
Gender [Count of Participants; unit: Participants]
  Female | 21
  Male | 15
Region of Enrollment [Number; unit: participants]
  Canada | 36

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response Rate (Defined as Partial or Complete Response as Defined by the RECIST Criteria)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 8 years
Measure: Number; unit: participants
Arm/Group | Treatment (Temsirolimus)
Number analyzed (Participants) | 36
participants | 2

2. Secondary Outcome: Stable Disease Rate Defined by RECIST Criteria
Description: Potential association between variables will be measured using Pearson correlation coefficients, chi-square tests, one- or two-sample t-tests or logistic regression analyses as appropriate. Ninety-five percent confidence intervals will be constructed and selected results will be illustrated using figures and plots.
Time Frame: Up to 8 years
Measure: Number; unit: participants
Arm/Group | Treatment (Temsirolimus)
Number analyzed (Participants) | 36
participants | 20

3. Secondary Outcome: Median Survival Time
Description: Computed using the Kaplan-Meier method.
Time Frame: 3
Population: Out of the 25 patients alive (in 2006 at time of publication)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Temsirolimus)
Number analyzed (Participants) | 25
months | 13.9 [2.8 to 22.6]

4. Secondary Outcome: Survival Rate
Description: Computed using the Kaplan-Meier method.
Time Frame: 1 year
Population: Out of the 25 patients alive as of Jan 2006
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Temsirolimus)
Number analyzed (Participants) | 25
percentage of participants | 71.5 [57.1 to 89.5]

5. Secondary Outcome: Response and Stable Disease
Description: Assessed using RECIST criteria.Patients that had Stable disease for 2 months
Time Frame: 2 months
Population: Number of patients that had stable disease for 2 months
Measure: Number; unit: patients
Arm/Group | Treatment (Temsirolimus)
Number analyzed (Participants) | 36
patients | 20

6. Secondary Outcome: Number of Temsirolimus Treatment Cycle Analyzed for Toxicity
Description: Safety and tolerability of treatment with Temsirolimus assessed using CTCAE v 3
Time Frame: Duration of participants treatment upto 16wks (4cycles) of treatment
Measure: Number; unit: treatment cycles
Arm/Group | Treatment (Temsirolimus)
Number analyzed (Participants) | 36
treatment cycles | 213

7. Secondary Outcome: Time to Progression
Time Frame: Up to 8 years
Population: At the time of publication, 5 patients were still on treatment and analysis was done on 31 patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Temsirolimus)
Number analyzed (Participants) | 31
months | 6.0 [3.7 to NA] — Not reached

ADVERSE EVENTS:
Arm/Group | Treatment (Temsirolimus)
Serious Adverse Events (participants affected / at risk) | 1/36
Other Adverse Events (participants affected / at risk) | 28/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Temsirolimus) (N=36)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Temsirolimus) (N=36)
Fatigue (General disorders) | 28
Hyperglycemia (Metabolism and nutrition disorders) | 25
rash / desquamation (Skin and subcutaneous tissue disorders) | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less